CLINICAL TRIAL: NCT05580601
Title: Haploidentical Donor Cytokine-Induced Memory-Like Natural Killer Cells (CIML-NK) for Relapsed & Refractory Acute Myeloid Leukemia (AML)
Brief Title: Cytokine-Induced Memory-Like Natural Killer Cells (CIML-NK) for Relapsed & Refractory Acute Myeloid Leukemia (AML)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0853
Record Dates: First submitted 2022-10-07; First posted 2022-10-14 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cytokine-Induced Memory-Like Natural Killer (CIML-NK) Cells (Experimental): The investigational cell product is a cytokine-induced memory-like natural killer cell preparation, derived from the recipient's haploidentical donor's apheresis product.
  Interventions: Drug: CIML-NK Cells

INTERVENTIONS:
Drug: CIML-NK Cells — The investigational cell product is a cytokine-induced memory-like natural killer cell preparation, derived from the recipient's haploidentical donor's apheresis product. At the time of infusion, the product is comprised of:
  * Cytokine-Induced Memory-Like NK cells (CIML-NK cells)
  * Human Serum Albumin
  * Plasmalyte
  The concentration and total cell number of CIML-NK cells in the product will vary based on the recipient body weight and the dose requested.

SUMMARY:
The objective of this study is to demonstrate that cytokine-induced memory-like natural killer cells can be generated from donor cells and infused safely into patients with relapsed or refractory acute myeloid leukemia (AML). A secondary objective is to assess efficacy of the CIML-NK cells in treating AML.

DETAILED DESCRIPTION:
The goal of treatment of relapsed or refractory acute myeloid leukemia (AML) is to achieve remission and proceed to hematopoietic stem cell transplant (HSCT). Unfortunately, standard protocols have limited success. In this study the investigators will identify patients with relapsed or refractory AML who are unlikely to benefit from standard chemotherapy protocols and do not qualify for, or do not wish to participate in, institutional chemotherapy trials. Peripheral blood from a related haploidentical donor will be collected for the isolation of natural killer (NK) cells. NK cells will be induced into a memory-like state using cytokine supplementation only. In this Phase I/II study, Patients will receive a lymphodepleting chemotherapy regimen, after which the cytokine-induced memory-like NK cells (CIML-NKs) will be infused. The primary study endpoint is the feasibility and safety of infusion of the cells. The secondary endpoints are efficacy, as measured by clinical response per standard CR/CRi criteria and ability to subsequently undergo allogeneic HSCT, and the persistence of memory-like NK cells in the blood as measured by flow cytometry.

ELIGIBILITY:
Inclusion Criteria:

* Of age ≥ 2 years of age at the time of study enrollment
* With AML diagnosed per 2016 WHO criteria (11)
* With relapsed or refractory AML in their bone marrow
* Refractory disease: Patients must have ≥ 5% blasts in the bone marrow after 2 courses of intensive induction treatment
* Relapsed disease: Patients must have ≥ 5% blasts in the bone marrow, or reappearance of blasts in the blood, within 6 months of initial CR
* With available haploidentical related donors. Donor specific antibody (DSA) testing will be done on the recipient prior to or upon enrollment.
* With performance level of ≥ 50% on Karnofsky scale for patients > 16 years of age and ≥ 50% on Lansky scale for patients ≤ 16 years of age

Exclusion Criteria:

* Disease: isolated central nervous system (CNS) disease, or isolated extramedullary disease, or diagnosis of acute promyelocytic leukemia (APML). Patients with extramedullary disease in combination with bone marrow disease are eligible for enrollment.
* Infectious Disease: Active uncontrolled infection
* Cardiac function: Systolic ejection fraction <45% by echocardiogram
* Pulmonary Function: Oxygen saturation <92% on room air
* Hepatic function: Total bilirubin > 2mg/dL, AST and ALT more than three times the upper limit of normal
* Concomitant medications: receiving either >10mg prednisone equivalent daily, or >0.5mg/kg prednisone equivalent daily, whichever is less
* Concomitant investigational treatments: receiving other investigational therapies
* Known allergy or hypersensitivity reaction to IL-2 injections
* Pregnant or breastfeeding women will not be entered on this study due to risks of fetal and teratogenic adverse events with lymphodepleting chemotherapy. Pregnancy tests must be obtained for female patients. Males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method while on study treatment and for six months following completion. Effective contraceptive methods include oral contraceptive pills, patches, or injections, intrauterine devices, having a tubal ligation, having a partner who has had a vasectomy, or not having sex.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-05-05 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Feasibility of infusion | 30 days
  Number of patients who receive CIML-NK infusion without grade 3-4 infusional toxicity events as assessed by CTCAE v5.0 divided by the number of patients enrolled.

SECONDARY OUTCOMES:
Clinical Response to CIML-NK Infusion | 30 days
  Clinical response to CIML-NK infusion assessed by bone marrow morphology per standard International Working Group CR/CRi criteria (Complete Remission (CR)
Persistence of CIML-NK cells in the recipients' peripheral blood | Assessed at day 7, 14, 21, 28
  Persistence of CIML-NK cells in the recipients' peripheral blood, assessed by flow cytometry
Proceed to Hematopoietic Stem Cell Transplant (HSCT) | 6 months
  Proportion of patients who are able to proceed to hematopoietic stem cell transplant

CONTACTS AND LOCATIONS:
Overall Officials: Zahra Hudda, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States